CLINICAL TRIAL: NCT07064005
Title: Brain Glutathione (GSH) Enrichment Through Gamma-glutamylcysteine (GGC) Supplementation in Early Parkinson's Disease Patients for Reduction of Extrapyramidal Motor Disturbances and Halting Cognition Decline: A Pilot Trial
Brief Title: Enrichment of Glutathione Using Gamma-glutamylcysteine Supplementation in Parkinson's Disease Patients.
Acronym: PDGSH
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pravat Mandal (Other)
Collaborators: Waste Connections Inc (Unknown)
Responsible Party: Sponsor-Investigator, Pravat Mandal, Research Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY24120097; 2001 (Other Grant/Funding Number: Waste Connections INC)
Record Dates: First submitted 2025-06-27; First posted 2025-07-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Parkinsons Disease (PD)
Keywords: Blood; Brain; MR Spectroscopy; GGC; Glutathione; Parkinsons disease; Oxidative stress; Brain Iron
MeSH Terms: conditions — Parkinson Disease | interventions — gamma-glutamylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gamma - Glutamylcysteine (Experimental): Patients will receive GGC tablet 400mg orally twice a day (morning and in the afternoon).
  Interventions: Drug: Gamma- glutamylcysteine

INTERVENTIONS:
Drug: Gamma- glutamylcysteine — 400 mg (two times) per day
  Other Names: GGC

SUMMARY:
This study is designed l to evaluate the effects of GGC oral supplementation in early Parkinson's disease (PD) patients. The main objectives of the study are to evaluate:

1. To study the enrichment of master antioxidant, glutathione (GSH) levels in brain and blood of these PD patients compared to baseline due to GGC supplementation.
2. To study the changes in motor function, cognitive skills in PD patients due to GGC oral supplementation
3. To study impact of GGC on gut health on the PD patients.

DETAILED DESCRIPTION:
This study will measure brain glutathione using non- invasive, state-of-the-art MEGA-PRESS pulse sequence in pre and post GGC supplementation after 12 months. The GSH level will also be measured in the blood in pre and post GGC supplementation. Brain and blood iron level will be measured in pre and post GGC supplementation.

The neuropsychological examination and motor function will be performed in pre and post GGC supplementation.

This study will provide the relation of brain GSH enrichment with motor performance.

Our study will also provide any possible correlation with reduction of dysbiosis of the gut microbiome with GSH enrichment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Parkinson's Disease diagnosis.
* Montreal Cognitive Assessment (MoCA) greater than or equal to 26.
* Age (50 to 80 years of age).
* Ability to read and write in English.

Exclusion Criteria:

* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments in the eyes, skin, or body.
* Subjects with claustrophobia.
* Patients with a clinical diagnosis of Parkinson's disease dementia or dementia with Lewy bodies.
* Subjects with a history of cancer.
* Subjects with active psychosis or delirium.
* Subjects with chronic kidney (creatinine > 1.5mg/dL) or liver disease (AST ≥ 1.5 ULN; ALT ≥ 1.5 ULN) within 30 days prior to enrolment.
* Subjects on antioxidant therapy (ashwagandha, gingko biloba or N-acetylcysteine) or illicit drug abuse/dependence (cocaine, heroin, marijuana, or fentanyl).
* Subjects with previous traumatic head injury.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-11-27 (Estimated)

PRIMARY OUTCOMES:
Changes in brain glutathione levels (mM) in people with Parkinson's Disease using Magnetic Resonance Spectroscopy compared to post-supplementation with GGC. | 12 months
  MEGA-PRESS is a non-invasive imaging technique, to detect various neurochemical (e.g., Glutathione) using 1H MR spectroscopy.
Changes in brain iron levels (ppb) in people with Parkinson's Disease using Magnetic Resonance Imaging between pre and post GGC supplementation. | 12 months
Changes in baseline blood iron levels(ng/μl) in people with Parkinson's Disease | 12 months
Changes in baseline blood glutathione levels (µmol/l) in people with Parkinson's Disease compared to post-supplementation with GGC | 12 months

SECONDARY OUTCOMES:
Monitor the change in the motor function using Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) pre and post GGC supplementation. | 12 months
  Scoring Method: Each section of the UPDRS is scored on a scale from 0 to 4.The total UPDRS score is calculated by summing the scores from each section, ranging from 0 (no disability) to 176 (severe disability).
  Interpretation: Higher scores indicates greater severity of symptoms.
Cognitive functions modulation- pre and post GGC supplementation using Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). | 12 months
  Interpretation: Higher scores indicate greater cognitive function.
Changes from baseline in the psychological distress using Brief Symptom Inventory (BSI-18) (self-report) in people with Parkinson's Disease. | 12 months
  Scoring Method: Each item is scored on a 0-4 scale, with the total score indicating the severity of distress. Interpretation: Higher total scores indicate greater severity of psychological distress.
Changes from baseline in the cognitive functions like memory, attention and decision-making using PROMIS Cognitive Function - Abilities-Short Form 8a (self-report) in people with Parkinson's Disease. | 12 months
  Scoring Method: Raw Score: 8-40 Interpretation: Lower scores on this measure indicate greater subjective cognitive difficulty.
Changes from baseline cognitive functions like attention, processing speed, and mental flexibility using Trail Making Test (TMT) A&B in people with Parkinson's Disease. | 12 months
  Scoring Method: The average scores are as follows: • Trail A - 29 seconds • Trail B - 75 seconds Interpretation: Higher scores indicate greater impairment

CONTACTS AND LOCATIONS:
Overall Officials: Pravat K Mandal, PHD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) collected during the trial, specifically data such as specimen type, relevant clinical characteristics based on primary and secondary outcome measures as reported in the summary results.
Supporting Information: CSR
Time Frame: The IPD report will be accessible starting 6 months after publication of the main results.
Access Criteria: Collaborating researchers with IRB approval or individuals listed on data use agreements may obtain data or specimens. The PI, Dr. Pravat K Mandal, University of Pittsburgh, mandalpk@pitt.edu, in collaboration with the research team, will review each request through email to ensure compliance with institutional policies, ethical standards, and any relevant data use agreements. All requests will be reviewed and responded to within 30 days.

REFERENCES:
- [Background] Dias V, Junn E, Mouradian MM. The role of oxidative stress in Parkinson's disease. J Parkinsons Dis. 2013;3(4):461-91. doi: 10.3233/JPD-130230. PMID 24252804
- [Background] Shukla D, Goel A, Mandal PK, Joon S, Punjabi K, Arora Y, Kumar R, Mehta VS, Singh P, Maroon JC, Bansal R, Sandal K, Roy RG, Samkaria A, Sharma S, Sandhilya S, Gaur S, Parvathi S, Joshi M. Glutathione Depletion and Concomitant Elevation of Susceptibility in Patients with Parkinson's Disease: State-of-the-Art MR Spectroscopy and Neuropsychological Study. ACS Chem Neurosci. 2023 Dec 20;14(24):4383-4394. doi: 10.1021/acschemneuro.3c00717. Epub 2023 Dec 5. PMID 38050970
- [Background] Mandal PK, Dwivedi D, Joon S, Goel A, Ahasan Z, Maroon JC, Singh P, Saxena R, Roy RG. Quantitation of Brain and Blood Glutathione and Iron in Healthy Age Groups Using Biophysical and In Vivo MR Spectroscopy: Potential Clinical Application. ACS Chem Neurosci. 2023 Jun 21;14(12):2375-2384. doi: 10.1021/acschemneuro.3c00168. Epub 2023 May 31. PMID 37257017